CLINICAL TRIAL: NCT03482414
Title: Improving Patient Motivation and Participation in Rehabilitation Program Through Social Games: A 3-arm Randomized Controlled Trial
Brief Title: Improving Patient Motivation and Participation in Rehabilitation Program Through Social Games
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: AWWA Rehab and Day Care Centre (Unknown)
Responsible Party: Principal Investigator, Wang Pan, Principal Investigator, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUSingapore_WP
Record Dates: First submitted 2018-02-01; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Stroke
Keywords: stroke; upper limb rehabilitation; neuro-rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: 3-arm randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- traditional wooden checkerboard (Active Comparator): upper limb training with traditional wooden checkerboard
  Interventions: Other: traditional wooden checkerboard
- gaming board with single-player games (Experimental): upper limb training with a LED-based interactive gaming board equipped with single-player games
  Interventions: Other: gaming board with single-player games
- gaming board with two-player games (Experimental): upper limb training with two LED-based interactive gaming boards equipped with two-player competitive games
  Interventions: Other: gaming board with two-player games

INTERVENTIONS:
Other: traditional wooden checkerboard — upper limb training with traditional wooden checkerboard
  Other Names: checkerboard for upper limb training
  Arms: traditional wooden checkerboard
Other: gaming board with single-player games — upper limb training with a LED-based interactive gaming board equipped with single-player games
  Other Names: interactive gaming board with single-player games
  Arms: gaming board with single-player games
Other: gaming board with two-player games — upper limb training with two LED-based interactive gaming boards equipped with two-player competitive games
  Other Names: interactive gaming board with two-player competitive games
  Arms: gaming board with two-player games

SUMMARY:
This 12-week randomized controlled trial involves two intervention groups (i.e., single-player game group, competition game group) and one control group (i.e., conventional checkerboard group). The main objective of this study is to examine the effects of game-based training on patient motivation, exercise duration, and functional outcomes in comparison with the control group.

DETAILED DESCRIPTION:
A 12-week three-arm randomized controlled trial was conducted to compare the effects between the single-player game, competitive game and a control group (i.e. conventional training) on the motivation, exercise duration and functional improvement in a rehabilitation program. A mix of quantitative method (i.e., questionnaire) and qualitative methods (i.e., interview and observation) were used. The outcome measurements were: (1) motivation: Intrinsic Motivation Inventory (IMI), (2) participation: exercise duration, (3) functional improvement: nine-hole peg test (NHPT) and box and block test (BBT), and (4) user feedback.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥65 years
2. Has neurological disorders (e.g. cerebrovascular accident) with the need of upper limb rehabilitation;
3. Able to stand or sit unsupported for 10 minutes;
4. Discharged from hospital and living in community;
5. Able to communicate either in English or Mandarin; and
6. Able to provide informed written consent.

Exclusion Criteria:

1. Has severe cognitive impairments (Mini-Mental State Examination (MMSE) score <10),
2. With serious cardiorespiratory conditions,
3. With capacity but do not wish to sign the consent form.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline motivation at 12 weeks | week 1, week 12
  Intrinsic Motivation Inventory (IMI) - psychological measurement of motivation questionnaire

SECONDARY OUTCOMES:
Change from baseline function of manual dexterity at 12 weeks | week 1, week 12
  Measuring gross manual dexterity Block and Box Test (BBT)
Change from baseline function of finger dexterity at 12 weeks | week 1, week 12
  Measuring finger dexterity with Nine-Hole Peg Test (NHPT)
Exercise duration | week 1 to week 12
  Overall exercise duration over12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pan Wang, Principal Investigator — National University of Singapore
Locations (1):
- Wang Pan, Singapore, Singapore - No State, Singapore

REFERENCES:
- [Background] McDonnell M. Action research arm test. Aust J Physiother. 2008;54(3):220. doi: 10.1016/s0004-9514(08)70034-5. No abstract available. PMID 18833688
- [Background] McAuley E, Duncan T, Tammen VV. Psychometric properties of the Intrinsic Motivation Inventory in a competitive sport setting: a confirmatory factor analysis. Res Q Exerc Sport. 1989 Mar;60(1):48-58. doi: 10.1080/02701367.1989.10607413. PMID 2489825
- [Background] Mathiowetz V, Volland G, Kashman N, Weber K. Adult norms for the Box and Block Test of manual dexterity. Am J Occup Ther. 1985 Jun;39(6):386-91. doi: 10.5014/ajot.39.6.386. PMID 3160243
- [Background] Oxford Grice K, Vogel KA, Le V, Mitchell A, Muniz S, Vollmer MA. Adult norms for a commercially available Nine Hole Peg Test for finger dexterity. Am J Occup Ther. 2003 Sep-Oct;57(5):570-3. doi: 10.5014/ajot.57.5.570. PMID 14527120
- [Background] Popovic MD, Kostic MD, Rodic SZ, Konstantinovic LM. Feedback-mediated upper extremities exercise: increasing patient motivation in poststroke rehabilitation. Biomed Res Int. 2014;2014:520374. doi: 10.1155/2014/520374. Epub 2014 Jun 2. PMID 24991557